CLINICAL TRIAL: NCT01998906
Title: A Randomized, Open-label Study of the Effect of Paclitaxel, Doxorubicin, and CMF Neoadjuvant Chemotherapy, With and Without Herceptin, on Tumor Response in Women With HER2-positive Breast Cancer
Brief Title: A Study of Herceptin (Trastuzumab) in Combination Chemotherapy in Women With Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO16432
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Results first posted 2014-10-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Doxorubicin; Paclitaxel

ARMS (3):
- HER-2+ Trastuzumab, Doxorubicin/Paclitaxel/CMF (Experimental): Participants with HER2 proto-oncogene positive breast cancer (HER2+) were treated with trastuzumab 8 milligrams per kilogram (mg/kg), intravenous (IV), on Day 1 of Cycle 1, followed by 6 mg/kg, IV, on Day 1 of Cycle 2 to up a maximum of Cycle 17. Participants also received doxorubicin 60 mg/ square meter (m^2), IV, and paclitaxel 150 mg/m^2, IV, on Day 1 of Cycles 1 through 3. Followed by paclitaxel 175 mg/m^2, IV, alone on Day 1 of Cycles 4 through 7. Participants also received CMF: cyclophosphamide 600 mg/m^2, IV; methotrexate 40 mg/m^2, IV; and 5-fluorouracil 600 mg/m^2, IV, on Day 1 of Cycles 8 through 10.
  Interventions: Drug: Trastuzumab; Drug: Doxorubicin; Drug: Paclitaxel; Drug: CMF
- HER-2+ Doxorubicin/Paclitaxel/CMF (Active Comparator): Participants with HER2 proto-oncogene positive breast cancer were treated with doxorubicin 60 mg/m^2, IV, and paclitaxel 150 mg/m^2, IV, on Day 1 of Cycles 1 through 3. Followed by paclitaxel 175 mg/m^2, IV, alone on Day 1 of Cycles 4 through 7. Participants also received CMF on Day 1 of Cycle 8 through 10.
  Interventions: Drug: Doxorubicin; Drug: Paclitaxel; Drug: CMF
- HER-2- Doxorubicin/Paclitaxel/CMF (Active Comparator): Participants with HER2 proto-oncogene negative breast cancer were treated with doxorubicin 60 mg/m^2, IV, and paclitaxel 150 mg/m^2, IV, on Day 1 of Cycles 1 through 3. Followed by paclitaxel 175 mg/m^2, IV, alone on Day 1 of Cycles 4 through 7. Participants also received CMF on Day 1 of Cycle 8 through 10.
  Interventions: Drug: Doxorubicin; Drug: Paclitaxel; Drug: CMF

INTERVENTIONS:
Drug: Trastuzumab — 8mg/kg IV on Day 1 of Cycle 1, followed by 6 mg/kg on Day 1 of Cycle 2 up a maximum of Cycle 17
  Other Names: Herceptin
  Arms: HER-2+ Trastuzumab, Doxorubicin/Paclitaxel/CMF
Drug: Doxorubicin — 60 mg/m2 IV on Day 1 of Cycles 1 through 3
Drug: Paclitaxel — 150 mg/m2 IV on Day 1 of Cycles 1 through 3, followed by 175 mg/m2 IV on Day 1 of Cycles 4 through 7
Drug: CMF — CMF: Cyclophosphamide (600 mg/m2 IV bolus), methotrexate (40 mg/m2 IV bolus), 5-fluorouracil (600 mg/m2 IV bolus) on Day 1 of Cycles 8 through 10

SUMMARY:
This study will assess the efficacy and safety of adding Herceptin to a paclitaxel-containing regimen followed by cyclophosphamide/methotrexate/fluorouracil (CMF) chemotherapy in women with locally advanced breast cancer and HER2/c-erbB-2 gene amplification. In a parallel observational study patients with HER2-negative disease will receive the same chemotherapy without Herceptin.

ELIGIBILITY:
Inclusion Criteria:

* female patients, >=18 years of age, with locally advanced breast cancer.

Exclusion Criteria:

* previous therapy for any invasive malignancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2002-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (28):
- Vienna, Austria
- München, Germany
- Italy (15):
  - San Giovanni Rotondo, Apulia
  - Bologna, Emilia-Romagna
  - Carpi, Emilia-Romagna
  - Udine, Friuli Venezia Giulia
  - Milan, Lombardy
  - Pavia, Lombardy
  - Varese, Lombardy
  - Sassari, Sardinia
  - Trento, Trentino-Alto Adige
  - Pisa, Tuscany
  - Bellunoi, Veneto
  - Castelfranco Veneto, Veneto
  - Mirano, Veneto
  - Santorso, Veneto
  - Vicenza, Veneto
- Lisbon, Portugal
- Russia (3):
  - Kazan'
  - Moscow
  - Saint Petersburg
- Spain (7):
  - Barcelona, Barcelona
  - Terrassa, Barcelona
  - Jerez de la Frontera, Cadiz
  - Donostia / San Sebastian, Guipuzcoa
  - Madrid, Madrid
  - Valencia, Valencia
  - Zaragoza, Zaragoza

RESULTS

PARTICIPANT FLOW:
Groups:
- HER2+ Trastuzumab/Doxorubicin/Paclitaxel/CMF (HER2+TC): Participants with human epidermal growth factor receptor 2 proto-oncogene positive (HER2+) breast cancer received treatment as follows:
  Cycles 1-3 (3-week cycles): trastuzumab 8 milligrams per kilogram (mg/kg), intravenously (IV) on Day 1 (Cycle 1 only; 6 mg/kg in Cycles 2 and 3), doxorubicin 60 mg/square meter (mg/m^2), IV, and paclitaxel 150 mg/m^2, IV, on Day 1 followed by 2 weeks off.
  Cycles 4-7 (3-week cycles): trastuzumab 6 mg/kg, IV, paclitaxel 175 mg/m^2, IV, on Day 1, followed by 2 weeks off.
  Cycles 8-10 (3-week cycles): trastuzumab 6 mg/kg, IV, on Day 1 and cyclophosphamide 600 mg/m^2, IV, methotrexate 40 mg/m^2, IV, and 5-fluorouracil 600 mg/m^2, IV, (collectively CMF) on Days 1 and 8, followed by 2 weeks off.
  Cycles 11-17 (3-week cycles): postoperatively, participants received trastuzumab 6 mg/kg IV on Day 1, followed by 2 weeks off for maximum of 17 overall cycles with trastuzumab. Adjuvant tamoxifen, 20 mg/day was administered for up to 5 years.
- HER2+ Doxorubicin/Paclitaxel/CMF (HER2+C): Participants with HER2+ breast cancer received treatment as follows:
  Cycles 1-3 (3-week cycles): doxorubicin 60 mg/m^2, IV and paclitaxel 150 mg/m^2, IV, on Day 1 followed by 2 weeks off.
  Cycles 4-7 (3-week cycles): paclitaxel 175 mg/m^2, IV, on Day 1, followed by 2 weeks off.
  Cycles 8-10 (3-week cycles): cyclophosphamide 600 mg/m^2, IV, methotrexate 40 mg/m^2, IV, and 5-fluorouracil 600 mg/m^2, IV, on Days 1 and 8, followed by 1 week off.
- HER2- Doxorubicin/Paclitaxel/CMF (HER2-C): Participants with human epidermal growth factor receptor proto-oncogene negative (HER2-) breast cancer received treatment as follows:
  Cycles 1-3 (3-week cycles): doxorubicin 60 mg/m^2, IV, and paclitaxel 150 mg/m^2, IV, on Day 1, followed by 2 weeks off.
  Cycles 4-7 (3-week cycles): paclitaxel 175 mg/m^2, IV, on Day 1, followed by 2 weeks off.
  Cycles 8-10 (3-week cycles): cyclophosphamide 600 mg/m^2, IV, methotrexate 40 mg/m^2, IV, and 5-fluorouracil 600 mg/m^2, IV, on Days 1 and 8, followed by 1 week off.
Period: Overall Study
Arm/Group | HER2+ Trastuzumab/Doxorubicin/Paclitaxel/CMF (HER2+TC) | HER2+ Doxorubicin/Paclitaxel/CMF (HER2+C) | HER2- Doxorubicin/Paclitaxel/CMF (HER2-C)
Started | 115 | 116 | 99
Completed | 1 | 2 | 1
Not Completed | 114 | 114 | 98
Not completed — Participants ongoing in follow-up | 77 | 60 | 58
Not completed — Death | 21 | 30 | 17
Not completed — Lack of Efficacy | 10 | 9 | 8
Not completed — Failure to return | 0 | 2 | 4
Not completed — Violation of Selection Criteria | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 4 | 3
Not completed — Administrative/Other | 2 | 1 | 3
Not completed — Other | 3 | 8 | 4

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who were randomized for the main study or registered for the observational parallel study and who received study medication at least once. Groups were analyzed as randomized/registered. Age was missing for 1 participant in the HER2+ TC treatment group.
Groups:
- HER2+ TC: Participants with HER2+ breast cancer received treatment as follows:
  Cycles 1-3 (3-week cycles): trastuzumab 8 mg/kg, IV on Day 1 (Cycle 1 only; 6 mg/kg in Cycles 2 and 3), doxorubicin 60 mg/m^2, IV, and paclitaxel 150 mg/m^2, IV, on Day 1 followed by 2 weeks off.
  Cycles 4-7 (3-week cycles): trastuzumab 6 mg/kg, IV, paclitaxel 175 mg/m^2, IV, on Day 1, followed by 2 weeks off.
  Cycles 8-10 (3-week cycles): trastuzumab 6 mg/kg, IV, on Day 1 and cyclophosphamide 600 mg/m^2, IV, methotrexate 40 mg/m^2, IV, and 5-fluorouracil 600 mg/m^2, IV, (collectively CMF) on Days 1 and 8, followed by 2 weeks off.
  Cycles 11-17 (3-week cycles): postoperatively, participants received trastuzumab 6 mg/kg IV on Day 1, followed by 2 weeks off for maximum of 17 overall cycles with trastuzumab. Adjuvant tamoxifen, 20 mg/day was administered for up to 5 years.
- HER2+ C: Participants with HER2+ breast cancer received treatment as follows:
  Cycles 1-3 (3-week cycles): doxorubicin 60 mg/m^2, IV and paclitaxel 150 mg/m^2, IV, on Day 1 followed by 2 weeks off.
  Cycles 4-7 (3-week cycles): paclitaxel 175 mg/m^2, IV, on Day 1, followed by 2 weeks off.
  Cycles 8-10 (3-week cycles): cyclophosphamide 600 mg/m^2, IV, methotrexate 40 mg/m^2, IV, and 5-fluorouracil 600 mg/m^2, IV, on Days 1 and 8, followed by 1 week off.
- HER2- C: Participants with HER2- breast cancer received treatment as follows:
  Cycles 1-3 (3-week cycles): doxorubicin 60 mg/m^2, IV, and paclitaxel 150 mg/m^2, IV, on Day 1, followed by 2 weeks off.
  Cycles 4-7 (3-week cycles): paclitaxel 175 mg/m^2, IV, on Day 1, followed by 2 weeks off.
  Cycles 8-10 (3-week cycles): cyclophosphamide 600 mg/m^2, IV, methotrexate 40 mg/m^2, IV, and 5-fluorouracil 600 mg/m^2, IV, on Days 1 and 8, followed by 1 week off.
- Total: Total of all reporting groups
Arm/Group | HER2+ TC | HER2+ C | HER2- C | Total
Number analyzed (Participants) | 115 | 112 | 99 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (9.78) | 52.3 (10.97) | 50.6 (10.46) | 51.0 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 112 | 99 | 326
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival (EFS) - Percentage of Participants With an Event
Description: EFS was defined as the time between randomization and date of documented occurrence of disease recurrence or progression (local, regional, distant or contralateral) or death due to any cause.
Time Frame: Baseline (BL), Presurgery: Day 1 (Cycles 1-7) and Days 1 and 8 (Cycles 8-10); Postsurgery: Day 1 (Cycles 1-17); every 6 months up to 60 months after last dose of study drug; yearly thereafter
Population: The full analysis set (FAS) included all participants who were randomized in the main study or registered in the parallel observational arm.
Measure: Number; unit: percentage of participants
Arm/Group | HER2+ TC | HER2+ C | HER2- C
Number analyzed (Participants) | 115 | 116 | 99
percentage of participants | 40.0 [47.7 to NA] | 50.9 [24.1 to NA] | 42.4 [57.7 to NA]

2. Secondary Outcome: Percentage of Participants With Breast Pathological Complete Response (bpCR)
Description: bpCR was defined as an absence of any invasive cancer cell of the primary tumor at the time of major surgery after neoadjuvant chemotherapy with and without trastuzumab.
Time Frame: BL, Day 1 of Cycles 1-10 (pre-surgery)
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HER2+ TC | HER2+ C | HER2- C
Number analyzed (Participants) | 115 | 116 | 99
percentage of participants | 44.3 [35.1 to 53.9] | 26.7 [18.9 to 35.7] | 19.2 [12.0 to 28.3]
Statistical Analysis 1: Comparison: HER2+ TC vs HER2+ C; Test type: Superiority or Other; p = 0.0051, Chi-squared; Mean Difference (Final Values) = 17.6, 95% CI 2-sided [5.0 to 30.2]

3. Secondary Outcome: Percentage of Participants With Total Pathological Complete Response (tpCR)
Description: tpCR was defined as a determination of bpCR and an absence of positive axillary nodes on pathology.
Time Frame: BL, Day 1 of Cycles 1-10 (pre-surgery)
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HER2+ TC | HER2+ C | HER2- C
Number analyzed (Participants) | 115 | 116 | 99
percentage of participants | 40.0 [31.0 to 49.6] | 20.7 [13.7 to 29.2] | 18.2 [11.1 to 27.2]
Statistical Analysis 1: Comparison: HER2+ TC vs HER2+ C; Test type: Superiority or Other; p = 0.0014, Chi-squared; Mean Difference (Final Values) = 19.3, 95% CI 2-sided [7.2 to 31.4]

4. Secondary Outcome: Percentage of Participants Achieving Either Complete Response (CR) or Partial Response (PR) According to Modified Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Assessments were made based on objective tumor measurements of the lesions as recorded in the case report form. In inflammatory cancer, progressive disease (PD) was defined as progression of any of the 2 signs of breast edema and erythema. In non-inflammatory cancer, PD was concluded if either the investigator judged the participant as having progressed at any time prior to surgery, or there was at least a 20% increase in the sum of target lesions (TLs), any new lesion, or clear progression of any nontarget lesion (NTLs). Clear progression of any NTL was defined as at least a 20% increase in the sum of NTLs compared to BL. PR was defined as at least a 30% decrease from BL in the sum of the longest diameter of TLs. CR was defined as no PD as assessed by the investigator and complete disappearance of all lesions.
Time Frame: BL, Presurgery: Day 1 of Cycles 1-10
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HER2+ TC | HER2+ C | HER2- C
Number analyzed (Participants) | 115 | 116 | 99
percentage of participants | 72.7 [63.4 to 80.8] | 66.4 [56.6 to 75.2] | 65.6 [55.2 to 75.0]
Statistical Analysis 1: Comparison: HER2+ TC vs HER2+ C; Test type: Superiority or Other; p = 0.3077, Chi-squared; Mean Difference (Final Values) = 6.4, 95% CI 2-sided [-6.4 to 19.1]

5. Secondary Outcome: Overall Survival (OS) - Percentage of Participants With an Event
Description: OS was defined as the time from the date of randomization to the date of the death due to any cause.
Time Frame: BL, Presurgery: Day 1 (Cycles 1-7) and Days 1 and 8 (Cycles 8-10); Postsurgery: Day 1 (Cycles 1-17); every 6 months up to 60 months after last dose of study drug; yearly thereafter
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | HER2+ TC | HER2+ C | HER2- C
Number analyzed (Participants) | 115 | 116 | 99
percentage of participants | 19.1 [NA to NA] | 28.4 [58.2 to NA] | 21.2 [NA to NA]

6. Primary Outcome: Event-Free Survival
Description: The median time, in months, between randomization and date of documented occurrence of an EFS event.
Time Frame: as for outcome 5
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Groups:
- HER2+ C: Participants with HER2+ breast cancer received doxorubicin, paclitaxel and CMF as follows:
  Cycles 1-3 (3-week cycles): doxorubicin 60 mg/m^2, IV and paclitaxel 150 mg/m^2, IV, on Day 1 followed by 2 weeks off.
  Cycles 4-7 (3-week cycles): paclitaxel 175 mg/m^2, IV, on Day 1, followed by 2 weeks off.
  Cycles 8-10 (3-week cycles): cyclophosphamide 600 mg/m^2, IV, methotrexate 40 mg/m^2, IV, and 5-fluorouracil 600 mg/m^2, IV, on Day 1, followed by 2 weeks off.
- HER2- C: Participants with HER2- breast cancer received doxorubicin, paclitaxel, and CMF as follows:
  Cycles 1-3 (3-week cycles): doxorubicin 60 mg/m^2, IV, and paclitaxel 150 mg/m^2, IV, on Day 1, followed by 2 weeks off.
  Cycles 4-7 (3-week cycles): paclitaxel 175 mg/m^2, IV, on Day 1, followed by 2 weeks off.
  Cycles 8-10 (3-week cycles): cyclophosphamide 600 mg/m^2, IV, methotrexate 40 mg/m^2, IV, and 5-fluorouracil 600 mg/m^2, IV, on Day 1, followed by 2 weeks off.
Arm/Group | HER2+ TC | HER2+ C | HER2- C
Number analyzed (Participants) | 115 | 116 | 99
months | NA [47.7 to NA] — Median and upper limit of the 95 percent (%) confidence interval (CI) could not be calculated due to an insufficient number of events at the time of analysis. | 43.6 [24.1 to NA] — Upper limit of the 95% CI could not be calculated due to an insufficient number of events at the time of analysis. | 64.5 [57.7 to NA] — Upper limit of the 95% CI could not be calculated due to an insufficient number of events at the time of analysis.
Statistical Analysis 1: Comparison: HER2+ TC vs HER2+ C; Test type: Superiority or Other; p = 0.0275, Log Rank; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.44 to 0.96]

7. Primary Outcome: Percentage of Participants Event Free at 1 Year
Time Frame: as for outcome 5
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HER2+ TC | HER2+ C | HER2- C
Number analyzed (Participants) | 115 | 116 | 99
percentage of participants | 89 [84 to 95] | 82 [74 to 89] | 80 [73 to 88]

8. Secondary Outcome: Overall Survival
Description: OS was defined as the time from the date of randomization to the date of the death due to any cause.
Time Frame: as for outcome 5
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HER2+ TC | HER2+ C | HER2- C
Number analyzed (Participants) | 115 | 116 | 99
months | NA [NA to NA] — Median and 95% CI could not be estimated at the time of data analysis due to the (expected) long survival duration of participants in the trial. | NA [58.2 to NA] — Median and upper limit of the 95% CI could not be estimated at the time of data analysis due to the (expected) long survival duration of participants in the trial. | NA [NA to NA] — Median and 95% CI could not be estimated at the time of data analysis due to the (expected) long survival duration of participants in the trial.
Statistical Analysis 1: Comparison: HER2+ TC vs HER2+ C; Test type: Superiority or Other; p = 0.0555, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.35 to 1.02]

9. Secondary Outcome: Percentage of Participants Surviving at 1 Year
Time Frame: as for outcome 5
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HER2+ TC | HER2+ C | HER2- C
Number analyzed (Participants) | 115 | 116 | 99
percentage of participants | 100 [100 to 100] | 99 [97 to 100] | 97 [93 to 100]

10. Primary Outcome: Percentage of Participants Event Free at 2 Years
Time Frame: as for outcome 5
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HER2+ TC | HER2+ C | HER2- C
Number analyzed (Participants) | 115 | 116 | 99
percentage of participants | 73 [64 to 81] | 61 [51 to 70] | 69 [60 to 78]

11. Secondary Outcome: Percentage of Participants Surviving at 2 Years
Time Frame: as for outcome 5
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HER2+ TC | HER2+ C | HER2- C
Number analyzed (Participants) | 115 | 116 | 99
percentage of participants | 95 [91 to 99] | 88 [82 to 94] | 90 [83 to 96]

12. Primary Outcome: Percentage of Participants Event Free at 3 Years
Time Frame: as for outcome 5
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HER2+ TC: Participants with HER2+ breast cancer received treatment as follows:
  Cycles 1-3 (3-week cycles): trastuzumab 8 mg/kg, IV on Day 1 (Cycle 1 only; 6 mg/kg in Cycles 2 and 3), doxorubicin 60 mg/m^2, IV, and paclitaxel 150 mg/m^2, IV, on Day 1 followed by 2 weeks off.
  Cycles 4-7 (3-week cycles): trastuzumab 6 mg/kg, IV, paclitaxel 175 mg/m^2, IV, on Day 1, followed by 2 weeks off.
  Cycles 8-10 (3-week cycles): trastuzumab 6 mg/kg, IV, cyclophosphamide 600 mg/m^2, IV, methotrexate 40 mg/m^2, IV, and 5-fluorouracil 600 mg/m^2, IV, (collectively CMF) on Day 1, followed by 2 weeks off.
  Cycles 11-17 (3-week cycles): postoperatively, participants received trastuzumab 6 mg/kg IV on Days 1 and 8, followed by 1 week off for maximum of 17 overall cycles with trastuzumab. Adjuvant tamoxifen, 20 mg/day was administered for up to 5 years.
Arm/Group | HER2+ TC | HER2+ C | HER2- C
Number analyzed (Participants) | 115 | 116 | 99
percentage of participants | 65 [56 to 74] | 52 [43 to 62] | 63 [53 to 72]

13. Secondary Outcome: Percentage of Participants Surviving at 3 Years
Time Frame: as for outcome 5
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HER2+ TC | HER2+ C | HER2- C
Number analyzed (Participants) | 115 | 116 | 99
percentage of participants | 85 [79 to 92] | 78 [70 to 86] | 85 [78 to 92]

ADVERSE EVENTS:
Time Frame: BL, presurgery treatment Cycles 1-10, postsurgery Cycles 1-17, every 6 months thereafter for up to 60 months; yearly thereafter until primary analysis has taken place, after which serious adverse events were collected only if treatment related.
Description: The safety analysis population included all participants randomized in the main study or registered in the parallel observational arm who received at least 1 dose of study medication. 20 participants in the HER2+C group crossed over to receive adjuvant trastuzumab after surgery; these participants were included in the HER+C group below.
Arm/Group | HER2+ TC | HER2+ C | HER2- C
Serious Adverse Events (participants affected / at risk) | 18/115 | 8/112 | 9/99
Other Adverse Events (participants affected / at risk) | 113/115 | 112/112 | 98/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HER2+ TC (N=115) | HER2+ C (N=112) | HER2- C (N=99)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 3 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Wound abscess (Infections and infestations) | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 2 | 0 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 3 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HER2+ TC (N=115) | HER2+ C (N=112) | HER2- C (N=99)
Angina pectoris (Cardiac disorders) | 6 | 5 | 0
Tachycardia (Cardiac disorders) | 6 | 6 | 1
Conjunctivitis (Eye disorders) | 34 | 22 | 7
Lacrimation increased (Eye disorders) | 15 | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 13 | 15 | 5
Abdominal pain lower (Gastrointestinal disorders) | 3 | 7 | 1
Abdominal pain upper (Gastrointestinal disorders) | 19 | 9 | 1
Constipation (Gastrointestinal disorders) | 15 | 20 | 11
Diarrhoea (Gastrointestinal disorders) | 35 | 32 | 18
Dyspepsia (Gastrointestinal disorders) | 9 | 3 | 7
Nausea (Gastrointestinal disorders) | 88 | 88 | 70
Stomatitis (Gastrointestinal disorders) | 46 | 44 | 21
Vomiting (Gastrointestinal disorders) | 54 | 52 | 36
Asthenia (General disorders) | 52 | 58 | 32
Chest pain (General disorders) | 7 | 9 | 2
Fatigue (General disorders) | 26 | 15 | 13
Influenza like illness (General disorders) | 26 | 26 | 0
Mucosal inflammation (General disorders) | 16 | 14 | 14
Oedema peripheral (General disorders) | 11 | 13 | 6
Pyrexia (General disorders) | 20 | 14 | 9
Hypersensitivity (Immune system disorders) | 1 | 4 | 5
Bronchitis (Infections and infestations) | 7 | 1 | 1
Cystitis (Infections and infestations) | 6 | 5 | 0
Influenza (Infections and infestations) | 14 | 23 | 5
Pharyngitis (Infections and infestations) | 8 | 1 | 1
Rhinitis (Infections and infestations) | 8 | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 7 | 3 | 7
Weight increased (Investigations) | 8 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 17 | 20 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 26 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 8 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 20 | 22 | 14
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 8 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 35 | 25 | 31
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 8 | 5
Dizziness (Nervous system disorders) | 9 | 10 | 2
Dysgeusia (Nervous system disorders) | 12 | 16 | 8
Headache (Nervous system disorders) | 14 | 16 | 8
Neuropathy peripheral (Nervous system disorders) | 25 | 26 | 5
Neurotoxicity (Nervous system disorders) | 6 | 4 | 6
Paraesthesia (Nervous system disorders) | 22 | 29 | 22
Peripheral sensory neuropathy (Nervous system disorders) | 16 | 17 | 23
Sensory disturbance (Nervous system disorders) | 10 | 10 | 11
Insomnia (Psychiatric disorders) | 7 | 6 | 4
Amenorrhoea (Reproductive system and breast disorders) | 15 | 13 | 14
Breast pain (Reproductive system and breast disorders) | 4 | 8 | 2
Menstruation irregular (Reproductive system and breast disorders) | 13 | 9 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 13 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 21 | 9 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 91 | 87 | 90
Alopecia totalis (Skin and subcutaneous tissue disorders) | 19 | 20 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 2 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 16 | 12 | 5
Nail disorder (Skin and subcutaneous tissue disorders) | 9 | 9 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 8 | 8 | 5
Hot flush (Vascular disorders) | 16 | 6 | 9
Hyperaemia (Vascular disorders) | 6 | 4 | 0
Hypertension (Vascular disorders) | 3 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.